CLINICAL TRIAL: NCT01509456
Title: The Effect of Potassium Bicarbonate on Bone and the Immune System During 21 Days of 6° Head- Down- Tilt Bedrest (HDT- Bedrest)
Brief Title: The Effect of Potassium Bicarbonate on Bone and Several Physiological Systems During Immobilisation
Acronym: NUC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DLR German Aerospace Center (Other)
Collaborators: University of Trieste (Other); University of Aarhus (Other); European Space Agency (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: AO-2004-068 (MAP)
Record Dates: First submitted 2011-07-04; First posted 2012-01-13 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Bone Diseases, Metabolic; Acid-Base Imbalance; Muscular Atrophy; Sprains and Strains; Protein Metabolism; Body Weight Changes; Cardiovascular Abnormalities
Keywords: bone metabolism; potassium bicarbonate; alkaline salt; acid base balance; bed rest
MeSH Terms: conditions — Bone Diseases, Metabolic; Acid-Base Imbalance; Muscular Atrophy; Sprains and Strains; Body Weight Changes; Cardiovascular Abnormalities | interventions — potassium bicarbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Potassium Bicarbonate (Active Comparator)
  Interventions: Dietary Supplement: Potassium Bicarbonate
- Control (No Intervention)

INTERVENTIONS:
Dietary Supplement: Potassium Bicarbonate — 90 mmol daily, effervescent tablets 30 mmol diluted in 200 ml tab water supplemented three times a day together with the main meals for 21 days of HDT- bedrest
  Arms: Potassium Bicarbonate

SUMMARY:
Mainly due to the absence of gravitational forces in weightlessness, astronauts suffer from an increased bone loss- negatively affecting health and vitality during a mission. The development of effective countermeasures to this loss includes many different aspects like sports but also nutrition.

Alkaline salts, abundant in fruits and vegetables, have shown to have positive effects on markers of bone turnover of postmenopausal women but also men and younger adults. With the current study the effects of a potassium bicarbonate supplementation added to a standardised, strictly controlled, definite diet of healthy, young men, should be verified within 21 days of 6°- HDT- Bedrest- the gold standard of simulating weightlessness within earthbound conditions.

DETAILED DESCRIPTION:
Astronauts in space suffer from an increased bone loss which is mainly related to the absence of gravitational forces. This increased bone reduction is accompanied by an higher concentration of calcium in urine and in this respect enhancing the risk of renal stones. Due to the fact, that bones´ regeneration does not occur rapidly even after returning to earth, astronauts face an increased risk of osteoporosis.

Nutritional factors such as a deficient intake of calcium, energy and fluid and the abundant intake of table salt exhibit additional negative effects on bone. Results of several studies consistently show the negative effects of acids on bone (increased bone loss). With respect to space missions of longer duration one big challenge is the development of countermeasures for the negative consequences of weightlessness on bone.

As not all needed experiments for the development of countermeasures can be conducted in space, simulation models of weightlessness such as 6° Head- Down- Tilt- Bedrest (HDT- Bedrest) have been implemented on earth, miming some physiological conditions of weightlessness such as unloading and immobilisation of the lower parts of the body and the fluid shift.

Alkaline salts, such as potassium bicarbonate (KHCO3), demonstrate positive effects on bone when being supplemented to postmenopausal women. Apart from the positive effects on markers of bone turnover, calcium concentration in urine could be reduced. Thus, the main aim of the present study was to reduce the immobilization induced bone resorption through an alkalizing effect of the alkaline salt KHCO3's supplementation during Head- Down- Tilt- Bedrest (HDT- Bedrest)-a leading simulation model of weightlessness.

The crossover designed study consisted of two parts of equal length (36 days)- 7 days of adaptation, 21 days of HDT- Bedrest, 6 days recovery and 2 days of long- term follow- up. Both study parts only differed in the HDT- period, where one group of the 8 healthy, young, male participating subjects was supplemented with 90 mmol KHCO3 daily (3 times a day 30 mmol KHCO3 diluted in 200 ml tab water, supplemented together with the main meals), while the other group only received 200 ml of tab water without any supplementation (Control group).

The measurements of bone formation markers as well as bone resorption markers in blood and urine supply insight into the influences of the supplementation on bone metabolism while blood gas analysis together with the pH- values of the 24h- urine point out the alkalising effects of KHCO3. Further physiological systems like protein and muscle metabolism, body weight and body composition, circulation and the neuro- vestibular system are simultaneously under investigation.

ELIGIBILITY:
Inclusion Criteria:

* healthy male subjects
* age: 20- 45
* weight 65- 85 kg
* height: 158- 190 cm
* BMI 20- 26 kg/m2
* no high performance sports
* non- smoking (minimum 6 months prior to study start)
* willing to complete both parts of the study
* presentation of social security and criminal record
* successful completion of medical and psychological screening
* signed informed consent

Exclusion Criteria:

* drugs- and alcohol abuse
* antiinflammatory drugs taken during the study
* vegetarianism, veganism
* migraine
* psychical illness in the past
* claustrophobia
* hiatal hernia
* gastroesophageal reflux
* diabetes mellitus
* Rheumatic disease
* muscle or joint disease
* disc prolapse
* orthostatic intolerance
* Hyperlipidaemia
* renal disease
* thyroid dysfunction
* hyperhomocysteinaemia
* hyper-/hypouremia
* hyper-/hypocalcemia
* anaemia
* hypoferremia
* Vitamin D deficiency
* deviation of blood gases from normal values (pH 7,38 - 7,42; pO2 79 - 98 mmHg; pCO2 34 - 45 mmHg; HCO3 20 - 28 mmol/l; Base excess ± 2 mmol/l)
* risk of thrombosis
* chronic back pain
* bone fracture within one year prior to study start
* bone mineral density 1,5 SD ≤ t-Score
* metal implants or other osteosynthesis material
* subject within another clinical trial within 2 months prior to study start
* any other status which according to the apprehension of the principal investigator leads to the exclusion of the subject

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2010-02; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
The reduction of the immobilisation induced bone loss by supplementing an alkaline salt (potassium bicarbonate) | 21 days of HDT- Bedrest

SECONDARY OUTCOMES:
Influence of KHCO3 on bone mass, bone mineral density and bone strength | 21 days of HDT- Bedrest
Determination of effects of KHCO3 on muscle strength, muscle power and muscle volume | 21 days of HDT- Bedrest
Determine the effects of KHCO3 on body composition and body weight | 21 days of HDT- Bedrest
Determine the effects of KHCO3 on the cardiovascular system | 21 days of HDT- Bedrest
Determine the effects of KHCO3 on the neuro- vestibular system | 21 days of HDT- Bedrest
Determination of effects of KHCO3 on protein and muscle turnover | 21 days of HDT- Bedrest

CONTACTS AND LOCATIONS:
Overall Officials: Francisca May, Dr., Principal Investigator — German Aerospace Centre, Institute of Aerospace Medicine (DLR)
Locations (1):
- German Aerospace Centre (DLR), Cologne, Germany

REFERENCES:
- [Derived] Frings-Meuthen P, Bernhardt G, Buehlmeier J, Baecker N, May F, Heer M. The negative effect of unloading exceeds the bone-sparing effect of alkaline supplementation: a bed rest study. Osteoporos Int. 2019 Feb;30(2):431-439. doi: 10.1007/s00198-018-4703-6. Epub 2018 Sep 25. PMID 30255228